CLINICAL TRIAL: NCT01468285
Title: A Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Pilot Study to Evaluate the Effect of Betahistine on Cerebral Blood Flow and Gait in Subjects at Risk of Falling
Brief Title: The CBF Study Evaluating the Effect of Betahistine on the Cerebral Blood Flow
Acronym: CBF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Products (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S108.4.104
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Gait or Balance Disorder Problems
Keywords: interventional,placebo controlled
MeSH Terms: interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment arm 1: betahistine dihydrochloride (Experimental)
  Interventions: Drug: betahistine dihydrochloride
- Treatment arm 2: placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: betahistine dihydrochloride — betahistine dihydrochloride 24 mg tablet b.i.d. six weeks treatment
  Other Names: Agiserc®
  Arms: Treatment arm 1: betahistine dihydrochloride
Other: placebo — placebo tablets b.i.d., six weeks treatment
  Arms: Treatment arm 2: placebo

SUMMARY:
Betahistine may provide benefit by enhancement of Cerebral Blood Flow (CBF). This placebo-controlled pharmacodynamic treatment study will primarily explore the effect of betahistine on cerebral blood flow measured by dynamic contrast-enhanced MRI imaging, in a patient population with MRI evidence of cerebrovascular compromise. Also it will be measured if CBF changes correlate with gait and cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with gait or balance disorder problems
2. Male and female subjects aged on 40 years and above.
3. Absence of known contraindications for betahistine treatment.
4. Currently not on betahistine (of any formulation) treatment for at least 45 days prior to inclusion in the study.
5. Subject consuming caffeinated or alcoholic beverages should have stable consumption throughout the study period.

Exclusion Criteria:

1. History of discontinuation of betahistine treatment (of any formulation) in the past due to lack of efficacy or side effects.
2. Subjects treated with antihistamines and monoamine oxidase (MAO) inhibitors 30 days prior to inclusion in the study.
3. Subjects with hypersensitivity to the active substance or to any of the excipients of the drug.
4. Phaeochromocytoma
5. Porphyria

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow (CBF) | 6 weeks
  To explore the sustained effect of betahistine on the cerebral blood flow (CBF) in the whole brain.

SECONDARY OUTCOMES:
Regional Cerebral Blood Flow (rCBF) | 6 weeks
  To explore the sustained effect of betahistine on the regional cerebral blood flow (rCBF) in pre-determined regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Kazei, MD, Study Director — Abbott
Locations (2):
- Singapore (2):
  - Site Reference ID/Investigator# 63545, Singapore
  - Site Reference ID/Investigator# 63544, Singapore